CLINICAL TRIAL: NCT05925283
Title: Clinical Study of Oral Midazolam Combined With Esketamine Administered Intranasally for Pediatric Preoperative Sedation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2023-03-105
Record Dates: First submitted 2023-06-12; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam; Esketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- midazolam (Placebo Comparator): Patients were assigned to receive oral midazolam 0.5mg.kg-1 approximately 30-40 minutes before surgery using a computer-generated random number table.
  Interventions: Drug: Midazolam
- esketamine (Experimental): Patients were assigned to receive intranasal esketamine 1mg/kg approximately 30-40 minutes before surgery using a computer-generated random number table.
  Interventions: Drug: Esketamine
- midazolam and esketamine (Experimental): Patients were assigned to receive intranasal esketamine 0.6mg/kg and oral midazolam 0.3mg.kg-1 approximately 30-40 minutes before surgery using a computer-generated random number table.
  Interventions: Drug: midazolam and esketamine

INTERVENTIONS:
Drug: Midazolam — oral midazolam 0.5mg.kg-1 approximately 30-40 minutes before surgery using a computer-generated random number table.
  Other Names: oral midazolam
  Arms: midazolam
Drug: Esketamine — intranasal esketamine 1mg/kg approximately 30-40 mins before surgery using a computer-generated random number table.
  Other Names: Intranasal esketamine
  Arms: esketamine
Drug: midazolam and esketamine — oral midazolam 0.3mg/kg and intranasal esketamine 0.6mg/kg approximately 30-40 mins before surgery using a computer-generated random number table.
  Other Names: combination with intranasal esketamine and oral midazolam
  Arms: midazolam and esketamine

SUMMARY:
Children are prone to anxiety and even fear before surgery, and such adverse emotions may not only lead to poor induction of anesthesia, but also increase the incidence of postoperative agitation and even lead to postoperative behavioral changes in children. There are many ways to relieve pediatric anxiety, including preoperative medication, games, and cartoons. Preoperative medication is the most commonly used method to relieve pediatric anxiety.The most commonly used pediatric preoperative sedation drugs are midazolam and esketamine.However, oral midazolam may not produce a sedative effect in 20-40% of patients. A good preoperative anxiety-reducing effect was seen in only 60-80% of cases.Therefore, this trial investigates whether the intranasal combination of esketamine with oral midazolam can produce better results than each of the two drugs alone. This will provide a reference for the selection of safe, reliable and appropriate preoperative sedation methods for pediatric patients and provide evidence-based support for comfort care.

DETAILED DESCRIPTION:
A trained member of the research team obtained a baseline The Modified Yale Preoperative Anxiety Scale(mYPAS) after obtaining consent. And corresponding study medication is administered about 30-40 minutes before the anesthesia induction.Vital signs were measured every 5 min after study medication administration.The sedation scores of the children were recorded with University of Michigan Sedation Scale (UMSS) every 10 minutes.The onset time of satisfactory sedation and parental separation anxiety scale was noted.Then recorded the degree of cooperation during inhalation anesthesia induction and recovery times.Moreover, recorded the pediatric anesthesia emergence delirium scale (PAED) during the recovery period.

ELIGIBILITY:
Inclusion Criteria:

1. with American Society of Anesthesiologists (ASA) physical status I or II；
2. aged 2-6 years；
3. children with weight for age within the normal range
4. were scheduled lower abdominal and perineal surgery with an expected operation time shorter than 30 minutes.

Exclusion Criteria:

1. Children who had gastrointestinal,Cardiovascular or endocrine dysfunction;
2. contraindication to preoperative sedation or had a known allergy or hypersensitive reaction to either esketamine or midazolam;
3. with any nasal pathology,organ dysfunction;
4. recently respiratory infection, mental disorder;
5. other reasons that researchers hold it is not appropriate to participate in this trial.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
The degree of cooperation during inhalation anesthesia induction | During inhalation anesthesia induction
  Induction Compliance Checklist range from 0 through 10,and lower scores indicate the higher degree of cooperation during inhalation anesthesia induction

SECONDARY OUTCOMES:
Anxiety before induction of anesthesia | Each 10 minutes during the forty minutes of preoperative period
  The Modified Yale Preoperative Anxiety Scale:
  The 22-item measure has five behavioural categories: activity, emotional expressivity, alertness and arousal, vocalizations, and interaction with parents. Total scores range from 23.33 through 100 with higher scores indicating greater anxiety.
The level of sedation | Each 10 minutes during the forty minutes of preoperative period
  University of Michigan Sedation Scale:
  0 -Awake/Alert
  1 -Minimally Sedated: Tired/sleepy, appropriate response to verbal conversation and/or sounds.
  2- Moderately Sedated: Somnolent/sleeping, easily aroused with light tactile stimulation.
  3 - Deeply Sedated: Deep sleep, arousable only with significant physical stimulation.
  4 - Unarousable.
  higher scores mean a higher levels of sedation.
Parental separation anxiety scale | During the preoperative period
  A four-point parental separation anxiety scale as follows:
  1. -Easy separation,
  2. -Whimpers, but is easily reassured, not clinging,
  3. - Cries and cannot be easily reassured, but not clinging to parents,
  4. - Crying and clinging to parents.
  The scores of 1 and 2 signified acceptable separation whereas scores of 3 and 4 were classified as difficult separation.
Recovery times | Within up to 30 minutes after child's first eye opening in the postoperative period
  The time from discontinuation of sevoflurane to the first open eye of the children and to achieve aldrete≥9
Pediatric anesthesia emergence delirium | Within up to 15-30 minutes after child's first eye opening in the postoperative period
  The pediatric anesthesia emergence delirium scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20.
  The degree of emergence delirium increased directly with the total score.pediatric anesthesia emergence delirium scale ≥12 at any time indicates presence of emergence delirium.
Number of children with adverse effects | Up to 24 hours including preoperative, intraoperative, and postoperative periods
  Number of children with adverse effects
  1. Bradycardia and/or hypotension need for hemodynamic support
  2. Desaturation is defined as Oxygen desaturation <90%
  3. Salivation
  4. Any adverse effects requiring interventions

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Xulin Zhang, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No